CLINICAL TRIAL: NCT02000505
Title: Comparison of the Quality of CPR by Lay Rescuers With and Without Telephone Instructions by a Simulated Rescue Coordination Center
Brief Title: Comparison of the Quality of CPR by Lay Rescuers With and Without Feedback Devices
Acronym: frequenz
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Stefan Braunecker, Anesthesiologist, Researcher, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-333
Record Dates: First submitted 2013-11-17; First posted 2013-12-04 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): 5 minutes chest-compression-only CPR, without any support
- PocketCPR (Experimental): 5 minutes chest-compression-only CPR, with support
  Interventions: Device: PocketCPR
- Metronome (Experimental): 5 minutes chest-compression-only CPR, with support
  Interventions: Device: Metronome
- 110bpm Song (Experimental): 5 minutes chest-compression-only CPR, with support
  Interventions: Device: 110bpm Song

INTERVENTIONS:
Device: PocketCPR — 5 minutes chest-compression-only CPR, using Zoll PocketCPR
  Arms: PocketCPR
Device: Metronome — 5 minutes chest-compression-only CPR, using a metronome
  Arms: Metronome
Device: 110bpm Song — 5 minutes chest-compression-only CPR, using a song with 110bpm for support
  Arms: 110bpm Song

SUMMARY:
Comparison of various methods to improve the quality of CPR

DETAILED DESCRIPTION:
Even for paramedics and emergency physicians, the resuscitation of patients with cardiac arrest remains a challenge. Previous studies have shown that the cardiac output varies widely even among professional helpers. This is especially due to some very different mean frequencies of cardiac compression wich vary from 60 to 160/min for paramedics. Aim of this study is to investigate whether the use of feedback-devices during cardiac-pulmonary resuscitation (CPR) can lead to an improvement of the cardiac output and may improve survival.

For this, we examine the impact of different feedback-methods on the frequence-variety on manikin by lay rescuers. Overall, we compare three different devices for feedback during CPR. The subjects for this study are lay rescuers who perform a 5 minute chest-compression-only CPR.

ELIGIBILITY:
Inclusion Criteria:

* lay rescuers
* >18 years
* <60 years

Exclusion Criteria:

* professional rescuers
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The average achieved cardiac output | after 5 minutes
  The main goal of the study is the average achieved cardiac output. Data acquisition is carried out on a resuscitation-manikin which can measure compression-rate (CR) and compression-depth (CD). The data are recorded by a computer during the CPR. To calculate the cardiac output, we multiply the average CR [1/min] with the average CD [mm] during the 5 min manikin-resuscitation. The thus obtained average cardiac-output (CO = CR x CD), measured in [mm/min], will be compared in each group.

SECONDARY OUTCOMES:
Constancy of the quality of chest-compressions | after 5 minutes
  Second objective of the study is the variation of the compression-rate and the compression-depth during the resuscitation. We compare the average compression-rate and compression-depth of the first 30 compressions and the last 30 compression of every participant. As a result, the average standard deviation in each group will be calculated. Afterward, the groups will be compared using the mean deviation of every group. The mean deviation will be measured in +/-[mm] for compression-depth and +/-[1/min] for compression rate.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Braunecker, MD, Principal Investigator — University Hospital Cologne; Jochen Hinkelbein, MD, Study Director — University Hospital Cologne
Locations (1):
- Uniklinik Köln, Cologne, Germany